CLINICAL TRIAL: NCT01005914
Title: Phase II Trial of the Addition of PEG-Asparaginase to the Hyper-CVAD Regimen in Adult Newly-Diagnosed Acute Lymphoblastic Leukemia
Brief Title: Pegaspargase and Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Increased rate of bacterial infections
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Brandon Hayes-Lattin, Brandon M. Hayes-Lattin, M.D., OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004913; OHSU-4913 (Other: OHSU IRB); ENZON-OHSU-4913 (Other: OHSU); CDR0000642363 (Other: NCI PDQ)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Leukemia
Keywords: adults; Philadelphia chromosome precursor ALL,; T-cell ALL; untreated ALL
MeSH Terms: conditions — Leukemia; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; Doxorubicin; Imatinib Mesylate; Methotrexate; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; pegaspargase; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental): Drug:cyclophosphamide Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3
  Drug:cytarabine Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4
  Drug:dexamethasone Day 1-4; 11-14: 40 mg daily
  Drug:doxorubicin hydrochloride Day 4: 50 mg/m2 IV over 2 hours
  Drug:imatinib mesylate 600 mg/day
  Drug:methotrexate Day 1: 1g/ m2 (200 mg/ m2load IV over 2 hours plus 800 mg/ m2 over 22 hours as an infusion
  Drug: methylprednisolone Day 1-3: 50mg IV BID
  Drug: pegaspargase Day 3/Day4: 2,500 IU/ m2 IV
  Drug: vincristine sulfate Day 4 & 11: 2 mg IV
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: imatinib mesylate; Drug: methotrexate; Drug: methylprednisolone; Drug: pegaspargase; Drug: vincristine sulfate

INTERVENTIONS:
Drug: cyclophosphamide — Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3
  Other Names: Cytoxan, Neosar, CTX
Drug: cytarabine — Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4
  Other Names: Cytosar-U, Ara-C, Arabinosylcytosine
Drug: dexamethasone — Day 1-4; 11-14: 40 mg daily
  Other Names: Decadron, DexPak, dex
Drug: doxorubicin hydrochloride — Day 4: 50 mg/m2 IV over 2 hours
  Other Names: Adriamycin RDF, Adriamycin PFS
Drug: imatinib mesylate — 600 mg/day
  Other Names: Gleevec, Glivec
Drug: methotrexate — Day 1: 1g/ m2 (200 mg/ m2load IV over 2 hours plus 800 mg/ m2 over 22 hours as an infusion
  Other Names: Trexall, Rheumatrex, MTX
Drug: methylprednisolone — Day 1-3: 50mg IV BID
  Other Names: Medrol, Depo-Medrol, Solu-Medrol
Drug: pegaspargase — Day 3/Day4: 2,500 IU/ m2 IV
  Other Names: Onscapar, PEG-L-asparaginase
Drug: vincristine sulfate — Day 4 & 11: 2 mg IV
  Other Names: Marqibo

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving pegaspargase together with combination chemotherapy and to see how well it works in treating patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the complete response rate in patients with newly diagnosed acute lymphoblastic leukemia treated with pegaspargase in combination with hyper-CVAD regimen comprising cyclophosphamide, dexamethasone, vincristine sulfate, doxorubicin hydrochloride, methotrexate, and cytarabine.
* To determine the safety and tolerability of this regimen in these patients.

Secondary

* To evaluate the progression-free survival and overall survival of patients treated with this regimen.
* To determine the half-life of pegaspargase when administered in combination with hyper-CVAD regimen.
* To monitor the development of neutralizing antibodies to pegaspargase when administered in combination with hyper-CVAD regimen.
* To assess minimal residual disease by flow cytometry at the end of courses 1A and 1B.

OUTLINE: This is a multicenter study.

* Hyper-CVAD regimen (courses 1, 3, 5, and 7): Patients receive cyclophosphamide IV over 2-3 hours twice daily on days 1-3, dexamethasone IV on days 1-4 and 11-14, methotrexate intrathecally (IT) on day 2, doxorubicin hydrochloride IV over 2 hours and pegaspargase IV over 1-2 hours on day 4, vincristine sulfate IV on days 4 and 11, and cytarabine IT on day 8.
* High-dose methotrexate/cytarabine regimen (courses 2, 4, 6, and 8): Patients receive methotrexate IV continuously over 24 hours on day 1, methylprednisolone IV twice daily on days 1-3, methotrexate IT on day 2, cytarabine IV over 2 hours twice daily on days 2 and 3, pegaspargase IV over 1-2 hours on day 3, and cytarabine IT on day 8.

Treatment repeats every 3-4 weeks for 8 courses in the absence of disease progression or unacceptable toxicity. Patients with Philadelphia chromosome-positive disease also receive oral imatinib mesylate daily beginning at diagnosis.

Patients who complete 8 courses of chemotherapy and are not candidates for hematopoietic stem cell transplantation receive maintenance therapy off study.

Blood samples are collected at baseline and periodically during study for pharmacokinetics and neutralizing antibody assays.

After completion of study therapy, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed (untreated) with Acute Lymphoblastic Leukemia based on a bone marrow examination unless there is a contraindication to having the test performed. This includes precursor-B ALL, precursor-T ALL, and Philadelphia chromosome positive ALL. For reference, see criteria by Center for International Blood and Marrow Transplant Research (CIBMTR).> 20% blasts on a bone marrow aspirate OR If a bone marrow aspirate is not obtained, the diagnosis of acute leukemia can be established by a pathologic diagnosis of acute leukemia on a bone marrow biopsy OR A complete blood count documenting the presence of at least 10,000 white blood cells (WBC)/μl and at least 20% circulating blasts
* Adults, 18 to 60 years of age.
* Women of child bearing potential (WOCBP) must be willing to use adequate contraception to avoid pregnancy for the duration of study participation.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Adequate renal function defined as: Serum creatinine ≤ 2.0 x upper limit normal (ULN) for institution
* Adequate hepatic function defined as:Total bilirubin ≤ 2.0 x ULN for institution Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 x ULN for institution
* Patient must have the ability to understand and the willingness to sign a written informed consent document. The patient and/or the patient's legally authorized guardian must acknowledge consent for treatment as a human subject on this study.

Exclusion Criteria:

* Mature B (Burkitt's) ALL will be excluded.
* An active malignancy other than ALL (with the exception of basal and/or squamous cell skin cancers and curatively treated carcinoma of the cervix) within 5 past years of study entry.
* Documented central nervous system (CNS) involvement with leukemia will be excluded. A diagnostic lumbar puncture will not be part of screening procedures.
* Severe pulmonary, renal, or hepatic disease not related to the patient's ALL will be excluded.
* Cardiac dysfunction as defined by:Myocardial infarction within the last 6 months of study entry, or Reduced left ventricular function with an ejection fraction ≤50% as measured by Multigated Acquisition (MUGA) scan or echocardiogram at study entry, Unstable angina, Unstable cardiac arrhythmias, New York Heart Association (NYHA) Class III or IV heart failure, Electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Known or suspected human immunodeficiency virus (HIV)-positive patients are excluded from the study because of possible risk of lethal infection when treated with marrow suppressive therapy.
* Any concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, etc.) or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Patients who have had chemotherapy or radiotherapy for ALL prior to entering the study will be excluded. Hydroxyurea and one dose of intravenous vincristine are allowed prior to registration for patient convenience. Prior steroid therapy is allowable, ≤5 days prior to the start of the regimen.
* Patients may not have received any other investigational agents within the last 30 days.
* WOCBP who are unwilling or unable to use an acceptable method of contraception for the entire study period. Pregnant or lactating women are excluded from this study because of possible risk to the fetus or infant. Women with a positive serum pregnancy test on enrollment or prior to study drug administration will be excluded.
* Men whose sexual partners are WOCBP, who are unwilling or unable to use an acceptable contraceptive method to avoid pregnancy of his partner for the entire study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Hayes-Lattin, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Drug:cyclophosphamide-Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3 Drug:cytarabine Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4 Drug:dexamethasone Day 1-4; 11-14: 40 mg daily Drug:doxorubicin hydrochloride Day 4: 50 mg/m2 IV over 2 hours Drug:imatinib mesylate 600 mg/day Drug:methotrexate Day 1: 1g/ m2 (200 mg/ m2load IV over 2 hours plus 800 mg/ m2 over 22 hours as an infusion Drug: methylprednisolone Day 1-3: 50mg IV BID Drug: pegaspargase Day 3/Day4: 2,500 IU/ m2 IV Drug: vincristine sulfate Day 4 & 11: 2 mg IV
  cyclophosphamide: Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3
  cytarabine: Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4
  dexamethasone: Day 1-4; 11-14: 40 mg daily
  doxorubicin hydrochloride: Day 4: 50 mg/m2 IV over 2 hours
  imatinib mesylate: 600 mg/day
  methotrexate: D
Period: Overall Study
Arm/Group | Group 1
Started | 11
Completed | 1
Not Completed | 10
Not completed — Adverse Event | 4
Not completed — Death | 4
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Outcome data was not collected due to early termination of the study due to safety concerns.
Groups:
- Group 1: Drug:cyclophosphamide Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3 Drug:cytarabine Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4 Drug:dexamethasone Day 1-4; 11-14: 40 mg daily
  Drug:doxorubicin hydrochloride Day 4: 50 mg/m2 IV over 2 hours
  Drug:imatinib mesylate 600 mg/day
  Drug:methotrexate Day 1: 1g/ m2 (200 mg/ m2load IV over 2 hours plus 800 mg/ m2 over 22 hours as an infusion
  Drug: methylprednisolone Day 1-3: 50mg IV BID
  Drug: pegaspargase Day 3/Day4: 2,500 IU/ m2 IV
  Drug: vincristine sulfate Day 4 & 11: 2 mg IV
  cyclophosphamide: Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3
  cytarabine: Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4
  dexamethasone: Day 1-4; 11-14: 40 mg daily
  doxorubicin hydrochloride: Day 4: 50 mg/m2 IV over 2 hours
  imatinib mesylate: 600 mg/day
  methotrexate: D
Arm/Group | Group 1
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.9 [22 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate After Course 1 of Pegaspargase When Administered in Combination With Hyper-CVAD Regimen
Description: The complete response rate after 1A cycle of a PEG-Asparaginase and hyper-CVAD combination regimen will be estimated, and an exact 95% confidence interval will be computed using a binomial distribution.
Time Frame: After day 4 of treatment
Population: Outcome data for this study was not collected due to early termination of the study due to safety concerns. Only one subject completed the study.
Groups:
- Group 1: Cy D1- 3: 300 m g/m2 IV- 6 doses, mesna 600 mg/ m2 /day continuous IV D 1-3, ARAC D 2 & 3: 3g/m2 IV q12 X 4, Dex D1-4; 11-14: 40 mg daily, doxorubicin hydrochloride D4: 50 mg/m2 IV, imatinib mesylate 600 mg/day, MTX D1: 1g/ m2 200 mg/ m2 load IV plus 800 mg/ m2, methylprednisolone D 1-3: 50mg IV BID, pegaspargase D3/D4: 2,500 IU/ m2 IV, vincristine sulfate D4 & 11: 2 mg IV, Cy: D 1- 3: 300 m g/m2 IV 6 doses plus mesna 600 mg/ m2 /day, continuous infusion D 1-3. ARAC D 2 & 3: 3g/m2 IV q12 X 4, dex: D 1-4; 11-14: 40 mg daily, doxorubicin hydrochloride: D 4: 50 mg/m2 IV, imatinib mesylate: 600 mg/day, MTX: D 1: 1g/ m2 200 mg/ m2load IV plus 800 mg/ m2 IV, methylprednisolone: D 1-3: 50mg IV BID, pegaspargase: D 3/D4: 2,500 IU/ m2 IV, vincristine sulfate: D 4 & 11: 2 mg IV, pharmacological study: C1A: pre-dose between Days 1 to 4, C1A: D11 or 12., C1A: D18 or 19, C 1A: D25 or 26, C1A: D32 or 33 C1B: pre-dose between D1-3, C1B: D1 or 11 C1B: D17 or 18, C1B: D24 or 25 C1B: D31 or 32
Arm/Group | Group 1
Number analyzed (Participants) | 0

2. Primary Outcome: Grade 3 and 4 Toxicity Associated With the Combination of Peg-Asparaginase and Hyper-CVAD Which Include: Allergic Reactions, Elevated Liver Enzymes, Hyperbilirubinemia, Hyperglycemia, Central Nervous System (CNS) Thrombosis, and Pancreatitis.
Time Frame: The assessment of safety will be based mainly on the frequency of adverse events
Population: as for outcome 1
Arm/Group | Group 1
Number analyzed (Participants) | 0

3. Secondary Outcome: 2-year Progression-free Survival
Time Frame: After completion of 8 cycles
Population: as for outcome 1
Arm/Group | Group 1
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Patients Who Achieve Complete Response or Partial Response After Courses 1 and 2
Time Frame: An interim analysis of safety is planned after the enrollment of 15 evaluable patients.
Population: as for outcome 1
Arm/Group | Group 1
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: At least every 6 months until death.
Population: as for outcome 1
Arm/Group | Group 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Minimal Residual Disease
Description: Cycle 1A: Days 1 through 14 Cycle 1B: Days 1 through 8, after the first 14 days of cycle 1A
Time Frame: End of cycles 1A and 1B
Population: as for outcome 1
Arm/Group | Group 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Half-life of Pegaspargase
Time Frame: The approximate t½ in adult patients is 5.73 days. The half-life is independent of the dose administered, disease status, renal or hepatic function, age, or gender.
Population: as for outcome 1
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All unexpected adverse events (AEs) related, probably related or possibly related to the study drug which are equal or greater than Grade 3 and serious adverse events (SAEs) were assessed within 30 to 42 days after the last dose of chemotherapy treatment (up to 9 months).
Description: Adverse events collected:
  1. Unexpected AEs (when type or severity isn't listed in Expected AE List)
  2. Deaths within 30 days of drug admin.
  3. Grade ≥ 3 (related to the following):
     * Allergic reactions
     * CNS thrombosis/embolism
     * Coagulopathy
     * Elevated AST, ALT
     * Hyperbilirubinemia
     * Hyperglycemia
     * Hypertriglyceridemia
     * Pancreatitis
Groups:
- Group 1: cyclophosphamide D1- 3: 300 m g/m2 IV 6 doses plus mesna 600 mg/ m2 /day cont. IV D1-3, cytarabine D2 & 3: 3g/m2 IV, dexD1-4; 11-14: 40 mg daily, doxorubicin hydrochloride D4: 50 mg/m2 IV
  Drug:imatinib mesylate 600 mg/day
  Drug:methotrexate Day 1: 1g/ m2 (200 mg/ m2load IV over 2 hours plus 800 mg/ m2 over 22 hours as an infusion
  Drug: methylprednisolone Day 1-3: 50mg IV BID
  Drug: pegaspargase Day 3/Day4: 2,500 IU/ m2 IV
  Drug: vincristine sulfate Day 4 & 11: 2 mg IV
  cyclophosphamide: Day 1- 3: 300 m g/m2 IV over 2-3 hours every 12 hours for 6 doses plus mesna 600 mg/ m2 /day continuous infusion Days 1-3
  cytarabine: Day 2 & 3: 3g/m2 IV over 2 hours q12 X 4
  dexamethasone: Day 1-4; 11-14: 40 mg daily
  doxorubicin hydrochloride: Day 4: 50 mg/m2 IV over 2 hours
  imatinib mesylate: 600 mg/day
  methotrexate: D
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 9/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=11)
Bacillus species sepsis with encephalitis (Infections and infestations) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
neutropenic fever (Blood and lymphatic system disorders) | 4 (7)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Septic shock (Infections and infestations) | 2 (2)
Pulmonary embolism (Vascular disorders) | 1 (1)
Death (General disorders) | 1 (1)
hypokalemia, hyponatremia (Blood and lymphatic system disorders) | 1 (2)
fungemia, staph bacteremia (Infections and infestations) | 1 (1)
gnr bacteremia (Infections and infestations) | 1 (1)
anaphylaxis (Immune system disorders) | 1 (1)
acute epiglottitis (Infections and infestations) | 1 (1)
klebsiella bacteremia (Infections and infestations) | 1 (1)
gastoenteritis (Gastrointestinal disorders) | 1 (1)
pneumonia (streptoccocus bacteremia) (Infections and infestations) | 1 (1)
lung infection (fungal) (Infections and infestations) | 1 (1)
alpha-hemolytic streptococcal bacteremia (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated early due to safety concerns. Only one subject completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes